CLINICAL TRIAL: NCT03428997
Title: Human Comedogenicity Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CO-171106085430-SACT
Record Dates: First submitted 2018-01-19; First posted 2018-02-12 (Actual); Results first posted 2019-08-02 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Comedogenicity
MeSH Terms: interventions — Skin Cream

STUDY DESIGN:
Intervention Model Description: The experimental lotion and negative control were both applied to test sites on each subjects back.
Who Masked: Investigator
Masking Description: The evaluator was blind to the placement of the interventions on the test sites.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Lotion (Experimental): Test sites were patched with the lotion F #13451-131.
  Interventions: Device: Lotion
- Negative Control (Other): Test sites were patched with undosed occlusive patch.
  Interventions: Other: Negative Control

INTERVENTIONS:
Device: Lotion — Formulated Lotion F# 13451-131 was applied on an occlusive patch and placed on a test site on each subjects back three times a week for four weeks.
  Arms: Lotion
Other: Negative Control — Control. An undosed occlusive patch was placed on a test site on each subjects back three times a week for four weeks.
  Arms: Negative Control

SUMMARY:
Testing comedogenicity potential of a device cream on humans.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* 18 to 45 years old.
* Individuals that are willing to provide written informed consent and are able to read, speak, write, and understand English.
* Individuals who are acne-prone with large pores on the back, or individuals who have a history of acne vulgaris on the face or back.
* Individuals who have had at least a 2-week rest period since participation in any previous clinical studies involving patch applications on the back.
* Individuals who are willing to avoid direct sun exposure on the back and use of tanning beds for the duration of the study.
* Generally, in good health based on medical history reported by the subject.
* Have generally healthy skin condition appropriate for study assessments
* Available for the entire study duration.
* Individuals who are willing to keep patch sites as dry as possible and refrain from swimming or soaking in a hot tub for the duration of the study (no showering/bathing restrictions).
* Willing to cooperate and follow instructions.
* Female subjects, not of child-bearing potential, must meet at least one of the following criteria:

Had a hysterectomy and/or bilateral oophorectomy, Be post-menopausal (amenorrhea for at least 1 year), Had a Tubal Ligation, Surgical sterilization (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy);

* Female subjects, of child-bearing potential, must agree to practice a medically acceptable form of birth control during the study and 30 days after study completion. Females must have used such birth control for at least 3 months prior to study start;
* Medically acceptable forms of birth control that may be used by the subject and/or his/her partner include:

Established use of hormonal methods of contraception (oral, injected, implanted, patch or vaginal ring).

Barrier methods of contraception with or without spermicide: condom or occlusive cap (diaphragm or cervical/vault caps), Intrauterine device (IUD) or intrauterine system (IUS), Surgical sterilization (e.g., in a monogamous relationship with male partner with vasectomy that has been confirmed effective by sperm count check, tubal occlusion, hysterectomy, bilateral salpingectomy). Abstinence from heterosexual intercourse: When this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception;

Exclusion Criteria:

* Individuals with known allergies or sensitivities to common topical skincare products, including adhesives and/or cyanoacrylate (super glue) or ingredients to the test materials for a specific test panel.
* Deprived from liberty by a judiciary or administrative decision.
* Having undergone organ excision (kidney, lung, spleen, and liver), an organ transplant, or a skull concussion with extended loss of consciousness within the last 5 years or with present symptoms and/or side effects.
* Individuals with self-reported UNCONTROLLED metabolic conditions, such as diabetes, hypertension, hyper/hypothyroidism, hypercholesterolemia, etc.
* Individuals with CONTROLLED health conditions may be excluded from the study at the discretion of the PI or designee:

Subjects with conditions that do not affect the skin, such as hypertension and hypercholesterolemia, could be enrolled when their health condition is managed through diet, medication, etc.

Subjects with conditions, which might affect the skin, such as hyper/hypothyroidism, diabetes must be excluded, regardless whether their health condition is controlled or not.

* Subjects who are taking medication for chronic conditions (e.g., insulin, antihistamines, steroidal and non-steroidal anti-inflammatory drugs, antibiotics, etc...) - exception could be made for hypercholesterolemia.
* Individuals with adult asthma and/or epilepsy.
* Skin diseases on tested sites (e.g., psoriasis, eczema, erythema, edema, scars, wounds, melanomas, etc.), which may influence the outcome of the study;

  -----Supplemental Consent During the eligibility screening, individuals who indicate that they have previously had eczema will be advised of the Koebner phenomenon, which refers to the appearance of these conditions either at the patch site or unrelated sites. If the individual chooses to participate in the study, 2 copies of a supplemental consent form will be signed by the subject (1 for the study files and 1 will be given to the subject).
* Subjects who are self-reported to be pregnant, lactating or planning to become pregnant; females of child-bearing potential who are unwilling or unable to use an acceptable method of contraception during the study.
* Male subjects who have a pregnant partner.
* Male subjects whose partner is planning to become pregnant during the study period or is unwilling or unable to use an acceptable method of contraception.
* Simultaneous participation in any other type of clinical study.
* An individual who has any condition which in the PI's judgment makes the candidate an inappropriate subject for study participation.
* Subjects who are related to those persons involved directly or indirectly with the conduct of this study (i.e., PI, sub-investigators, study coordinators, other site personnel, employees of the Sponsor subsidiaries, contractors of the Sponsor, and the families of each).
* Individuals with a condition or situation which, in the PI's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.
* Individual viewed by the PI as not being able to complete the study.
* Subjects who are planning to use any new personal care products (e.g. makeup) or are planning to change existing brands during the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-02-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stephens and Associates, Richardson, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lotion and Negative Control: The Formulation Lotion F#13541-131 on an occlusive patch and the undosed occlusive patch (negative control) were each applied to a test site on each subject's back three times a week for four weeks.
Period: Overall Study
Arm/Group | Lotion and Negative Control
Started | 24
Completed | 16
Not Completed | 8
Not completed — Sponsor decision. | 1
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: Only subjects that completed the study per-protocol are included in the analysis.Each subject had each treatment patched on their back
Arm/Group | Lotion and Negative Control
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.8 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Microcomedone Score of Follicular Biopsies
Description: Grades for irritations/reactions were The following 5-point global assessment scale was used to grade the follicular biopsies for microcomedones: 0 None (0% No microcomedones) 0.5 Slight (1-24% Smallish horny masses)
  1. Mild (25-49% Smallish horny masses)
  2. Moderate (50-74% Moderately sized horny masses)
  3. Severe (75-100% Larger globoid microcomedones)
Time Frame: 28 days
Population: All study participants received both the test product and a negative control following a randomization.
Measure: Mean (Standard Deviation); unit: microcomedone score
Units Other Than Participants: Test Site
Groups:
- Lotion: The Formulation Lotion F#13541-131 on an occlusive patch was applied to a test site on each subject's back three times a week for four weeks.
- Negative Control: Undosed occlusive patch (negative control) was applied to a test site on each subject's back three times a week for four weeks.
Arm/Group | Lotion | Negative Control
Number analyzed (Participants) | 16 | 16
Number analyzed (Test Site) | 16 | 16
microcomedone score | 0.84 (0.51) | 0.97 (0.56)
Statistical Analysis 1: Comparison: Lotion; Testing hypothesis is that the mean score is equal between the compared treatments; Test type: Equivalence — Mixed-effects model, where the test material/negative control is a fixed effect and the subject is a random effect; p = 0.274, 2-sided t-test; Mean Difference (Final Values) = -0.12, Standard Error of Mean 0.11

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: All of the Adverse Events recorded during the study were related to test material sites.
Groups:
- Negative Control: The undosed occlusive patch (negative control) was applied to a test site on each subjects back three times a week for four weeks.
Arm/Group | Lotion | Negative Control
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 4/24 | 0/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lotion (N=24) | Negative Control (N=24)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Cracking/Fissures/Dryness/Scabbing (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Edema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pustule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vessicles (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator (PI) will provide Sponsor with at least sixty (60) days to review any Publication. No Publication that incorporates Sponsor Confidential Information will be submitted for publication without Sponsor's prior written consent. If requested in writing, the PI withholds such Publication for up to an additional sixty (60) days to allow for filing of a patent application.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT03428997/Prot_SAP_000.pdf